CLINICAL TRIAL: NCT05555979
Title: Qualitative, Cross-sectional Observational Study Exploring the Experience of Patients Prescribed Venetoclax+Rituximab or Bruton's Tyrosine Kinase Inhibitors for Chronic Lymphocytic Leukaemia in Clinical Practice in the UK
Brief Title: A Study to Assess Change in Patient Experience in Adult Participants With Chronic Lymphocytic Leukemia (CLL) Receiving Oral Venetoclax Tablets + Intravenous Rituximab or Bruton's Tyrosine Kinase Inhibitors Tablets in the United Kingdom
Acronym: ELECTRIC
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P23-486
Record Dates: First submitted 2022-09-23; First posted 2022-09-27 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Chronic Lymphocytic Leukemia
Keywords: Chronic Lymphocytic Leukemia; Rituximab; Bruton's Tyrosine Kinase Inhibitor; Venetoclax; Venclexta; Venclyxto; ABT-199; Cancer
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Chronic Lymphocytic Leukemia (CLL) Participants: Participants treated with venetoclax+rituximab or bruton's tyrosine kinase inhibitors in accordance with approved local label.

SUMMARY:
Chronic lymphocytic leukemia (CLL), a form of Non-Hodgkin's Lymphoma, is the most common type of leukemia in adults, affecting approximately 3,800 people in the UK each year. This study will evaluate the patient experience of CLL in adult participants who are prescribed venetoclax+rituximab or Bruton's tyrosine kinase inhibitors in the United Kingdom (UK).

Venetoclax+rituximab is a drug approved to treat CLL. Study participants will receive venetoclax+rituximab as prescribed by their study doctor in accordance with approved local label. Adult participants prescribed venetoclax+rituximab or Bruton's tyrosine kinase inhibitors will be enrolled. Around 140 participants will be enrolled in the study in approximately 10 sites in the UK.

Participants will receive venetoclax tablets to be taken by mouth and rituximab intravenous (IV) injection according to the approved local label.

There is expected to be no additional burden for participants in this trial. All study visits will occur during routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed diagnosis of chronic lymphocytic leukemia (CLL) (as defined by 2008 Modified International Workshop for Chronic Lymphocytic Leukemia National Cancer Institute Working Group (IWCLL NCI-WG) Guidelines).
* Has relapsed/refractory (R/R) disease having received only 1 prior line of treatment, which must have been a chemotherapy or chemoimmunotherapy treatment.
* Has treatment experience with venetoclax+rituximab (Ven+R) or bruton's tyrosine kinase inhibitor (BTKi)s that meets the criteria for inclusion described in the protocol, for which recruitment targets have not yet been met.

Exclusion Criteria:

* Previously treated with a BTKi, a BCL-2 inhibitor or other investigational agents.
* Has any other medical condition or disorder that, in the opinion of the site investigator or study director, could compromise participant's ability to give written informed consent and/or prevent or interfere with his or her ability to comply with study procedures and provide meaningful information about his or her CLL experience.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with second-line (2L) chronic lymphocytic leukemia (CLL) treated with venetoclax+rituximab or bruton's tyrosine kinase inhibitors per approved local label in the United Kingdom.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2022-12-14 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-04-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with a Change in Chronic Lymphocytic Leukemia (CLL) Symptoms | Day 1
  Number of participants who report a change in CLL symptoms through qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (10):
- United Kingdom (10):
  - Barts Health NHS Trust /ID# 252717, London, London, City of
  - Norfolk and Norwich University Hospitals NHS Foundation Trust /ID# 252720, Norwich, Norfolk
  - Nottingham City Hospital /ID# 252716, Nottingham, Nottinghamshire
  - Oxford University Hospitals NHS Foundation Trust /ID# 252715, Oxford, Oxfordshire
  - University Hospitals Sussex NHS Foundation Trust /ID# 252672, Worthing, West Sussex
  - University Hospitals of Leicester NHS Trust /ID# 252719, Leicester
  - The Royal Marsden NHS Foundation Trust /ID# 252655, London
  - Portsmouth Hospitals University NHS Trust /ID# 252722, Portsmouth
  - Sunderland Royal Hospital /ID# 252495, Sunderland
  - Taunton and Somerset NHS Foundation Trust /ID# 252721, Taunton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Clinical Study Report Synopsis — https://www.abbvieclinicaltrials.com/study/?id=P23-486#additional-resources-section